CLINICAL TRIAL: NCT06615323
Title: The Effect of Polyphonic Lullaby and Pish Pish Sound on Sleep Transition and Sleep Duration in Newborns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sevgi Beyazgül (Other)
Responsible Party: Sponsor-Investigator, Sevgi Beyazgül, midwife, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/239
Record Dates: First submitted 2024-09-22; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Newborn; Vitality
Keywords: newborn; Polyphonic Lullaby; Pish Pish Sound; Sleep

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Polyphonic Lullaby Group (Experimental): After discharge, mothers will be asked to listen to the Dandini Dandini Dastana lullaby by singer Mircan Kaya, which they downloaded from the YouTube application, from a distance of one meter (away from the baby's head to minimize radioactive effects) and by turning the phone to airplane mode just before sleep. In case of active sleep transition (signs of sleep transition such as slowing down muscle movements and closing eyes), the polyphonic lullaby volume will be gradually reduced. The polyphonic lullaby will be lowered to 55 decibels for the first 5 minutes after falling asleep and then to 25 decibels and then turned off. In order to reduce the effect of confounding factors, mothers in the polyphonic lullaby group who used another assistive method (breastfeeding/rocking to sleep) to put their babies to sleep will be excluded from the scope of the study.
  Interventions: Behavioral: Polyphonic Lullaby Group
- Pish Pish Sound Group (Experimental): After discharge, mothers will be asked to turn on the Piş Piş sound downloaded from the YouTube application and listen to it from a distance of one meter (away from the baby's head to minimize radioactive effects) and by turning the phone to airplane mode just before sleep. In case of active sleep (signs of sleep transition such as slowing down muscle movements and closing eyes), the piş piş sound will be gradually reduced. The polyphonic lullaby played will be at a volume level of 55 decibels for the first 5 minutes after falling asleep, then reduced to 25 decibels and then turned off. In order to reduce the effect of confounding factors, mothers in the piş piş sound group who use another assistive method (breastfeeding/rocking to sleep) to put their babies to sleep will be excluded from the scope of the research.
  Interventions: Other: Pish Pish Sound Group
- Model Group (No Intervention): The mothers in the control group will be given general sleep education on ensuring sleep hygiene before discharge, and brochures containing information on ensuring sleep hygiene will be distributed, and no other application will be made. In order to reduce the effect of confounding factors, the mothers in the control group will be asked at each interview whether they used any assistive methods to facilitate the transition to sleep, and newborns in the control group who were determined to use piş piş sounds or polyphonic lullabies will be excluded from the scope of the study.

INTERVENTIONS:
Behavioral: Polyphonic Lullaby Group — After discharge, mothers will be asked to play the Dandini Dandini Dastana lullaby by vocal artist Mircan Kaya, which they downloaded from the YouTube application, and listen to it from a distance of one meter (away from the baby's head to minimize radioactive effects) and by switching the phone to airplane mode just before sleep. In the event of active sleep (signs of sleep transition such as slowing down muscle movements and closing eyes), the polyphonic lullaby volume will be gradually reduced. The polyphonic lullaby will be played at a volume level of 55 decibels for the first 5 minutes after falling asleep, then reduced to 25 decibels and then turned off. In order to reduce the effects of confounding factors, mothers in the polyphonic lullaby group who use another assistive method (breastfeeding/rocking to sleep) to put their babies to sleep will be excluded from the study.
  Arms: Polyphonic Lullaby Group
Other: Pish Pish Sound Group — After discharge, mothers will be asked to turn on the Piş Piş sound downloaded from the YouTube application and listen to it from a distance of one meter (away from the baby's head to minimize radioactive effects) and by turning the phone to airplane mode just before sleep. In case of active sleep (signs of sleep transition such as slowing down muscle movements and closing eyes), the piş piş sound will be gradually reduced. The polyphonic lullaby played will be at a volume level of 55 decibels for the first 5 minutes after falling asleep, then reduced to 25 decibels and then turned off. In order to reduce the effect of confounding factors, mothers in the piş piş sound group who use another assistive method (breastfeeding/rocking to sleep) to put their babies to sleep will be excluded from the scope of the research.
  Arms: Pish Pish Sound Group

SUMMARY:
Sleep is the cornerstone of early development. Adequate sleep in children is important for proper growth, development and the child's health. Sleep is a dynamic process that develops and matures rapidly, especially in the first few years of life, from infancy to early adolescence. Daily sleep duration decreases with age, starting from the newborn period. At birth, babies show a sleep process that is compatible with their mothers' circadian rhythm. Newborns usually wake up in line with their nutritional needs and have short transitional sleep periods. At approximately 10-12 weeks of age, the first signs of circadian rhythm begin to develop and become apparent with increased sleep during the night. It has been reported that music positively affects mother-infant bonding, reduces babies' stress and creates positive physiological and behavioral changes. In a study examining mothers' views and practices on singing lullabies, it was seen that 87.6% of mothers said that singing lullabies soothes their children and prepares them for sleep, 88.3% prefer to sing lullabies before going to sleep while preparing their children for sleep, and 66.2% sing lullabies. Therefore, it is thought that the research will fill this gap in newborns.

DETAILED DESCRIPTION:
Sleep is the cornerstone of early development. At approximately 10-12 weeks of age, the first signs of the circadian rhythm begin to develop and become evident with increased nighttime sleep. The change in the total 24-hour sleep duration decreases as the baby grows, gradually adapting to the circadian sleep rhythm. Daily sleep duration in newborns decreases to 16-17 hours, 14-15 hours at 16 weeks of age, and 13-14 hours at 6 months of age. As the baby grows, the need for daytime sleep decreases, resulting in a shift towards more nighttime sleep patterns. In recent years, studies examining the effects of music, especially on newborns, have increased. Music is a complex auditory stimulus consisting of various components such as melody, rhythm, timbre, and harmony. When adults listen to music, these components are perceived as a phenomenological whole, but they are processed separately through a complex dual cortical and subcortical regions. Since the adult human brain does not have a single musical center, the neural substrates supporting musical perception and production vary depending on the musical task. Neuroimaging studies in neonates or infants have reported inconsistent results regarding cortical activation in response to musical stimuli. While two studies showed weak bilateral responses to musical stimuli, results from a functional magnetic resonance imaging (fMRI) study used to measure brain activity in 1- to 3-day-old neonates hearing excerpts of Western tone music and modified versions of the same excerpts suggest that the infant brain shows hemispheric specialization in right-lateralized auditory cortex activity for processing music in the early postnatal hours, and that the neural architecture underlying music processing in neonates is sensitive to changes in tone key as well as differences in consonance and dissonance. It has been found that infants can maintain distinct memory traces for polyphonic music and show a high preference for polyphonic music from 3 months onwards. Marie and Trainor (2014) hypothesize that this high-volume advantage may be mediated at the level of the auditory nerve at birth. In general, the presence of immature mismatch negativity (MMN) occurs when there is an occasional change or deviant stimulus in a continuing standard stimulus sequence. Again, this more complex MMN-like response to polyphonic stimuli has been reported to have a longer developmental trajectory than the MMN elicited by a single tone stimulus. Early musical involvement is very important for the auditory system, which mostly matures in the first 6 months after birth. Polyphonic lullabies, known in the literature as polyphony consisting of sounds or music, are music played especially during the rapid development period (0-4 years) of infants and children. When the literature was examined, no randomized controlled studies were found that revealed the effects of polyphonic lullabies and piş piş sounds on the transition to sleep and sleep duration in healthy newborns. It was thought that the research results would provide strong evidence to support the development of approaches to improving sleep in newborns.

ELIGIBILITY:
Inclusion Criteria:

For newborns)

* Being healthy
* Being between 37th and 42nd weeks of gestation
* Being between 2500-4000 kg at birth
* Being exclusively breastfed for the first 3 months
* Not having a hearing problem detected by the newborn hearing test Criteria for inclusion in the study (For mothers)
* Not working for the first three months after birth
* Not having any known chronic physical or mental problems
* Not having any known sleep problems
* Being literate
* Being able to communicate in Turkish

Exclusion Criteria:

Exclusion criteria from the study (For newborns)

* Having a congenital anomaly
* Having a history of being in the neonatal intensive care unit
* Having any health problems
* Those who switched to mixed or formula feeding during the follow-up period

Exclusion criteria from the study (For newborns)

* Those who develop any disease in the newborn (convulsion, upper respiratory tract infection, urinary tract infection, etc.)
* Newborns in the experimental group who were not exposed to polyphonic lullaby/piş piş sounds for two consecutive days within 3 months and for a total of 5 days (Source.. I could not find a source here, lullaby studies conducted on preterm babies, if you want, I can add from those sources)
* Newborns who did not fill out a regular weekly sleep diary
* Newborns who were put to sleep by other sleep initiation methods such as breastfeeding or shaking to sleep other than the specified methods (polyphonic lullaby/piş piş sounds) will be excluded from the study.

Ages: 0 Days to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Mother and baby information form | Must be taken 5 minutes before work.
  It consists of a total of 22 questions developed by the researcher and his consultant based on literature, to determine the sociodemographic and descriptive characteristics that may affect the sleep pattern of babies. Before the data collection form is applied, it will be sent to experts in the field and expert opinions will be obtained.

SECONDARY OUTCOMES:
Extended BISQ Infant Short Sleep Questionnaire | Must be taken 10 minutes before work.
  The expanded version of the "Infant Short Sleep Questionnaire" is a questionnaire developed by Sadeh in 2004 to screen for parenting practices, daytime and nighttime routines, sleep problems based on parental responses, and sleep environment during early childhood (0-36 months). The questionnaire has 13 items based on parental reports of the infant or toddler's sleep patterns. In addition, there are 4 items related to the sleep environment and 5 items assessing parents' perception of sleep problems.

OTHER OUTCOMES:
Sleep Diary | twice a week immediately after the procedure
  A sleep diary was prepared by the researcher and his consultant in line with the literature so that the mothers could answer the questions in the BISQ questionnaire regarding sleep patterns as closely as possible to the truth: the time they started their bedtime routine, the time they went to bed, the number of times they woke up at night, the time they stayed awake at night, the longest sleep time spent without waking up at night, the total sleep time at night, and the number of daytime sleeps/naps.
Infant Colic Scale | Must be taken 15 minutes before work.
  The items of the infant colic scale were evaluated on a 6-point Likert scale. Scale items were rated with a Likert-type scoring system ranging from 1 to 6. The rating was made from 1 (strongly disagree) to 6 (strongly agree). Negative questions were reverse coded to ensure consistency in the interpretation of scores.